CLINICAL TRIAL: NCT07373054
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes in the Treatment of Androgenic Alopecia: A Prospective, Randomized, Controlled Clinical Trial
Brief Title: Umbilical Cord Mesenchymal Stem Cell-Derived Exosomes in the Treatment of Androgenic Alopecia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, ChenXiaosong, professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025KY611
Record Dates: First submitted 2025-12-30; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Androgenic Alopecia
Keywords: Androgenic Alopecia; stem cell; exosome
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Minoxidil Treatment Group (Active Comparator)
  Interventions: Drug: Topical Minoxidil
- Combination Treatment Group (Traditional) (Active Comparator)
  Interventions: Procedure: Electric Microneedling; Biological: Traditional Exosome Lyophilized Powder
- Combination Treatment Group (Innovative) (Experimental)
  Interventions: Procedure: Electric Microneedling; Biological: Innovative Exosome Lyophilized Powder

INTERVENTIONS:
Drug: Topical Minoxidil — Following the standard treatment protocol, subjects were instructed to topically apply 1 mL of 5% minoxidil twice daily until the completion of the 3-month treatment course. Self-recorded usage of minoxidil was documented in a daily log, which was reviewed by the investigators during each treatment visit.
  Arms: Minoxidil Treatment Group
Procedure: Electric Microneedling — Performed with a needle length of ~1.2 mm (adjusted to scalp thickness) at 100-200 Hz. The procedure is conducted in sections (e.g., forehead, vertex, temporal regions) until mild pinpoint bleeding (indicating dermal stimulation) is achieved.
  Arms: Combination Treatment Group (Innovative); Combination Treatment Group (Traditional)
Biological: Traditional Exosome Lyophilized Powder — A solution of exosomes (3 mL) prepared using the traditional purification process, for topical application after microneedling.
  Arms: Combination Treatment Group (Traditional)
Biological: Innovative Exosome Lyophilized Powder — A solution of exosomes (3 mL) prepared using a novel purification process with an inner-outer bilayer membrane lyoprotection system, for topical application after microneedling.
  Arms: Combination Treatment Group (Innovative)

SUMMARY:
Androgenic Alopecia(AGA) is a highly prevalent condition for which existing pharmacological and surgical interventions present limitations and side effects, creating a clinical need for safer and more effective therapies. In response, human umbilical cord mesenchymal stem cell-derived exosomes (hUCMSC-Exos) have emerged as a cell-free therapeutic strategy. Characterized by their rich bioactive components, absence of tumorigenic risk, and high safety profile, hUCMSC-Exos represent a promising approach for hair regeneration. This study aims to evaluate the safety and efficacy of hUCMSC-Exos combined with automated microneedle delivery for treating AGA. By utilizing innovative lyophilization technology to maintain exosomal bioactivity and employing precision microneedle systems for enhanced delivery, this research seeks to provide a new generation solution for androgenic alopecia treatment.

DETAILED DESCRIPTION:
Androgenic Alopecia (AGA) is a prevalent hereditary condition with significant limitations in current treatment options. Pharmacological therapies are often associated with gender-specific restrictions and adverse effects including sexual dysfunction and hypertrichosis, while surgical and immunotherapeutic approaches face challenges of high cost, limited efficacy, and potential complications. These shortcomings highlight the urgent clinical need for safer and more effective treatment strategies. Human umbilical cord mesenchymal stem cell-derived exosomes (hUCMSC-Exos), nano-scale vesicles measuring 30-150 nm in diameter, present a promising alternative. Enriched with bioactive components including proteins and lipids, these cell-free structures demonstrate no proliferative capacity, tumorigenic risk, or significant cytotoxicity, offering a superior safety profile compared to conventional stem cell therapies. This study employs an innovative "dual-layer membrane lyophilization system" that maintains exosomal bioactivity while enabling room temperature storage and transportation through optimized freeze-drying and reconstitution processes.

To address transdermal delivery challenges, the research utilizes an automated microneedle system that overcomes the limitations of traditional injection and roller microneedle methods in achieving uniform penetration and depth control. This advanced delivery platform ensures precise, consistent, and efficient exosomal permeation into scalp tissues.This study aims to evaluate the safety and efficacy of the combined approach of hUCMSC-Exos and automated microneedle delivery for treating AGA. By integrating innovative lyophilization technology with precision delivery, this research seeks to establish a new generation therapeutic solution for androgenic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 to 60 years (inclusive), in good general health.
* Clinical diagnosis of androgenetic alopecia (AGA) according to the 2023 Chinese Clinical Practice Guideline: Diagnosis and Treatment of Androgenetic Alopecia, with a disease duration of less than 5 years and a Hamilton-Norwood scale classification of stage II to IV at the screening visit.
* Able to fully understand the study's content, procedures, potential benefits, and risks, and willing to provide written informed consent prior to any study-specific procedures.
* Agrees to comply with the study protocol and refrain from using any other treatments for alopecia for the duration of the study.

Exclusion Criteria:

* Unwilling or unable to provide written informed consent.
* History of any malignancy within the past 5 years (except for adequately treated non-scalp basal cell carcinoma or squamous cell carcinoma in situ).
* Hypotension (blood pressure < 90/60 mmHg) documented within 1 month prior to screening, or uncontrolled hypertension within 3 months prior to screening (defined as failure to achieve a target of < 140/90 mmHg while on a stable regimen of at least two antihypertensive medications).
* Known history of any systemic disease that may affect hair growth or confound study assessments (e.g., HIV infection, connective tissue disease, inflammatory bowel disease, hypothyroidism, iron deficiency anemia, malnutrition, syphilis).
* Known history of other forms of non-androgenetic alopecia (e.g., diffuse alopecia, alopecia areata, cicatricial alopecia).
* History of major organ dysfunction, significant autoimmune disease, or immunodeficiency.
* Known coagulation disorders, current use of anticoagulant or antiplatelet therapy (except low-dose aspirin), thrombophilia, or inherited bleeding disorders.
* Treatment with chemotherapy, cytotoxic drugs, scalp radiation, or laser/surgical hair restoration within 12 months prior to screening.
* History of hair transplantation, or need for long-term use of wigs, hairpieces, or hair bonding agents during the trial.
* History of severe or multiple drug allergies, atopy, known allergy to local anesthetics, or planned desensitization therapy during the study period.
* Presence of any active dermatological condition in the target scalp area that could interfere with evaluation (e.g., infection, seborrheic dermatitis, psoriasis, eczema, folliculitis, open wounds, scars, or atrophy).
* Participation in another interventional clinical trial within 4 weeks prior to screening (except for non-interventional studies or participants who only signed the informed consent form without receiving any investigational product).
* Any other medical or psychiatric condition that, in the judgment of the investigator, would compromise the subject's safety, compliance, or suitability for study participation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Hair Density in the Alopecia Area | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Trichoscopic hair count (hairs/cm²) in a fixed 1 cm² frontal/vertex scalp area.
Mean Change in Hair Shaft Diameter | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  The diameter of at least 20 randomly selected terminal hairs in the alopecia area will be measured using trichoscopy with integrated measurement software, and the mean value will be calculated,Unit of measure: micrometer (μm).
Vellus-to-Terminal Hair Ratio | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Within a standardized alopecia area , vellus hairs (diameter < 30 μm) and terminal hairs (diameter ≥ 30 μm) will be counted separately via trichoscopy,Their ratio will be calculated. This is a dimensionless value reported as a ratio (e.g., 0.5) or a percentage (e.g., vellus hair proportion of 50%).
Photographic Hair Density Score | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Standardized photographs (90-degree vertex and 45-degree frontal views) are taken under fixed conditions. A trained, blinded rater will assign a score based on a predefined photographic scale that correlates with hair density (e.g., 1=Sparse to 5=Dense).

SECONDARY OUTCOMES:
Physician Global Assessment | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Hair loss severity was assessed using the Hamilton-Norwood Classification Scale. It classifies male androgenetic alopecia into ordered categorical stages (I through VII) with recognized variant patterns (e.g., types IIA, IIIA, IVA, VIA). The scale's minimum defined stage is Stage I, representing minimal to no frontotemporal recession. The maximum defined stage is Stage VII, characterized by the most advanced presentation of fusion of the frontotemporal and vertex regions of alopecia, with only a narrow, posteriorly situated horseshoe-shaped band of residual parietal and occipital hair. Evaluations were independently performed by two physicians from the department. In cases of significant discrepancy between the two assessors, a third physician was consulted. The final result was derived from the two most concordant assessments.
Patient Satisfaction Evaluation | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Patient satisfaction was evaluated using a self-reported satisfaction scale. The scale categories were: Very Satisfied (improvement ≥ 75%), Satisfied (improvement 50% to 75%), Neutral (improvement 25% to 49%), and Dissatisfied (improvement ≤ 25%). The satisfaction rate was calculated as follows: (Number of Very Satisfied + Number of Satisfied) / Total number of patients × 100%.
Adverse Events Monitoring | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Adverse events, including but not limited to erythema, burning, pruritus, dryness, irritation, hyperpigmentation, edema, hypertrophic scarring, skin ulceration, and infection, were monitored.
Visual Analog Scale (VAS) for Pain | Within one week prior to treatment initiation, and at Weeks 4, 12, and 24 after the first treatment
  Pain was assessed using the Visual Analog Scale (VAS). A linear scale marked from 0 to 10 was used, where the "0" end was labeled "No Pain" and the "10" end was labeled "Worst Pain Imaginable." Patients were instructed to mark on the line corresponding to their subjective pain level, allowing for a quantitative assessment of pain intensity. The VAS scoring criteria were as follows:0: No Pain；1-3: Mild Pain；4-6: Moderate Pain；7-9: Severe Pain；10: Worst Pain Imaginable。

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Union Hospital of Fujian Medical University, Fuzhou, Fujian, China